CLINICAL TRIAL: NCT05525208
Title: Observer-Blind, Randomized, Controlled Study of Immunogenicity and Safety of SARS-Cov-2 Protein Subunit Recombinant Vaccine (Bio Farma) as a Booster Dose Against COVID-19 in Adults 18 Years of Age and Older
Brief Title: Booster Study of COVID-19 Protein Subunit Recombinant Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Universitas Padjadjaran (Other); Udayana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CoV2-Booster-0222
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; healthy population; Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Vaccine candidate and active comparator are masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Primary dose of inactivated (Sinovac®) vaccine (1) (Experimental): Subject who had received a complete primary dose of inactivated (Sinovac®) vaccine
  Interventions: Biological: SARS-CoV-2 subunit protein recombinant vaccine
- Primary dose of mRNA (Pfizer®) vaccine (1) (Experimental): Subject who had received a complete primary dose of mRNA (Pfizer®) vaccine
  Interventions: Biological: SARS-CoV-2 subunit protein recombinant vaccine
- Primary dose of Viral Vector (AstraZeneca®) vaccine (1) (Experimental): Subject who had received a complete primary dose of viral vector (AstraZeneca®) vaccine
  Interventions: Biological: SARS-CoV-2 subunit protein recombinant vaccine
- Primary dose of inactivated (Sinovac®) vaccine (2) (Experimental): Subject who had received a complete primary dose of inactivated (Sinovac®) vaccine
  Interventions: Biological: Active Comparator
- Primary dose of mRNA (Pfizer®) vaccine (2) (Experimental): Subject who had received a complete primary dose of mRNA (Pfizer®) vaccine
  Interventions: Biological: Active Comparator
- Primary dose of Viral Vector (AstraZeneca®) vaccine (2) (Experimental): Subject who had received a complete primary dose of viral vector (AstraZeneca®) vaccine
  Interventions: Biological: Active Comparator

INTERVENTIONS:
Biological: SARS-CoV-2 subunit protein recombinant vaccine — SARS-CoV-2 RBD subunit recombinant protein, manufactured by PT. Bio Farma
  Arms: Primary dose of Viral Vector (AstraZeneca®) vaccine (1); Primary dose of inactivated (Sinovac®) vaccine (1); Primary dose of mRNA (Pfizer®) vaccine (1)
Biological: Active Comparator — The Pfizer-BioNTech® COVID-19 vaccine or BNT162b2, is an mRNA vaccine encoding a P2 mutant spike protein (PS 2) and formulated as an RNA-lipid nanoparticle of nucleoside-modified mRNA (modRNA).
  Arms: Primary dose of Viral Vector (AstraZeneca®) vaccine (2); Primary dose of inactivated (Sinovac®) vaccine (2); Primary dose of mRNA (Pfizer®) vaccine (2)

SUMMARY:
Observer-blind, randomized, active-controlled prospective intervention study of Immunogenicity & Safety of SARS-Cov-2 Protein Subunit Recombinant Vaccine (Bio Farma) as a Booster Dose Against COVID-19 in Adults 18 Years of Age and Older.

DETAILED DESCRIPTION:
This trial is observer-blind, randomized, prospective intervention study. In this study 900 subjects who had received complete primary doses of authorized/approved inactivated (Sinovac®), mRNA (Pfizer®), or viral vector (AstraZeneca®) COVID-19 vaccine and willing to participate in the booster study by signing the consent form, will be involved in this trial.

Subject will be divided into six groups, each 150 subjects per arm who had received a complete primary dose of inactivated (Sinovac®) vaccine, mRNA (Pfizer®) vaccine, or viral vector (AstraZeneca®) vaccine will receive one booster dose of SARS-CoV-2 subunit protein recombinant vaccine or active control.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy adults 18 years of age and older.
2. Subjects who have previously received complete primary series of authorized/approved inactivated (Sinovac®), mRNA (Pfizer®), or viral vector COVID-19 vaccine (AstraZeneca®) with the last dose administered a minimum of 6 months prior to inclusion but not longer than 12 months prior to inclusion.
3. Subjects have been informed properly regarding the study and signed the informed consent form.
4. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial.
2. Subject who has received booster dose of COVID-19 vaccine.
3. Subject who has history of COVID-19 in the last 3 months (based on anamnesis or other examinations).
4. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. Women who are pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
6. History of asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
7. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
8. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
9. Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
10. Subjects who have history of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome.
11. Subjects receive any vaccination (other than COVID-19 vaccine) within 1 month before and after IP immunization.
12. Subjects plan to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the candidate vaccine | 14 days after booster vaccination
  Geometric Mean Titer (GMT) and GMT ratio of neutralizing antibody to the SARS-CoV-2

SECONDARY OUTCOMES:
Seropositive rate of the candidate vaccine | Baseline, 14 days and 6 months after booster vaccination
  Seropositive rate of neutralizing antibody
Seroconversion rate of the candidate vaccine | Baseline and 14 days after booster vaccination
  Seroconversion rate of neutralizing antibody
Seropositive rate and GMT of candidate vaccine | Baseline, 14 days, and 6 months after booster vaccination
  Seropositive rate and GMT of candidate vaccine
Seroconversion rate of the candidate vaccine | baseline and 14 days after booster vaccination
  Seroconversion rate of IgG antibody (RBD)
Comparison of immunogenicity between candidate vaccine and control group | Baseline, 14 days, and 6 months after booster vaccination
  Comparison of GMT, seroconversion rate, seropositive rate of neutralizing antibody and IgG antibody (RBD) between candidate vaccine and control group
Safety of the candidate vaccine | 28 days after booster vaccination
  Percentage of subjects with solicited and unsolicited Adverse Events (AE)
Serious Adverse Event (SAE) of the vaccine | 6 months after booster vaccination
  Percentage of subjects with at least 1 SAE

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, Prof, MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran
Locations (2):
- Indonesia (2):
  - Faculty of Medicine Universitas Udayana, Denpasar, Bali
  - Faculty of Medicine Universitas Padjadjaran, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No